CLINICAL TRIAL: NCT02865096
Title: The Correlation of Women's Sexual Health and Marijuana Use
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Becky Lynn, MD, MD, St. Louis University
Other Study IDs: 26860
Record Dates: First submitted 2016-08-04; First posted 2016-08-12 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Women's Sexual Health

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is attempting to determine whether there is any effect (worsening or improvement of sexual function) after marijuana consumption. Both users and non users of marijuana will be given the opportunity to participate by completing a questionnaire.

DETAILED DESCRIPTION:
Marijuana is the most commonly used illicit drug (19.8 million past-month users) according to the 2013 National Survey on Drug Use and Health (NSDUH).

There is a current movement towards the legalization of marijuana in various states and there are numerous claims of potential uses in medicine.

The internet is rich with nonscientific, non-evidence based information regarding the effects of marijuana on the sex lives of women. However, surprisingly little scientific research has been done on it.

Cannabis use and sexual function Endocannabinoids, which are structurally similar to cannabis (marijuana) help regulate a number of motivated behaviors and emotional states, including sexual function. There are a variety of ways that cannabinoids interact with the hormones and neurotransmitters that affect sexual behavior. This interaction has not been clearly elucidated but studies in rats have helped to clarify the relationship between cannabinoids and the hormones and neurotransmitters that affect sexual behavior.

In male rats, administration of tetrahydrocannabinol (THC, the psychoactive compound in marijuana) reduced sexual motivation. In female rats, the relationship between THC and sexual behavior is less clear. found that giving female rats a low dose of THC increased their receptivity to copulation. However a high dose interfered with receptivity, also found that THC stimulated receptivity and increased proceptivity ("courting behavior") in female hamsters.

Lopez et al found that in rats, giving a cannabinoid receptor blocker, increased sexual motivation during the estrous cycle. They then found that ovariectomized rats given a cannabinoid receptor agonist, had reduced sexual motivation. When exogenous estrogen and progesterone were given, this effect was attenuated.

The exact mechanism by which THC affects sexual function in women is unknown. It is known that THC and the hypothalamic-pituitary-gonadal (HPG) axis, which controls the sex hormones, interact with eachother. Acute administration of THC has been shown to inhibit LH and PRL secretion from the anterior pituitary in males and females. In females, high dose of THC can interfere with estrous and menstrual cycle timing and can delay or prevent ovulation. Cannabinoids inhibit or interfere with activity of the HPG axis and reduce secretion of several hormones which tend to have an inhibitory impact on sexual behavior.

It is known that dopamine is a key prosexual modulator in normal excitatory female sexual function. It is also known that the major effects of THC in the central nervous system are mediated by cannabinoid receptors. These receptors have been shown to enhance dopamine (Lazenka et al, 2015), which may be another pathway by which marijuana affects sexual function.

Human studies are limited. Questioned regular male and female marijuana users about their opinions regarding changes in the sexual experience when using marijuana. They found that when marijuana affects the sexual experience, it affects it positively. Marijuana did appear to increase desire mildly and enhances the quality of orgasm.

There are several links between THC and hormonal and neurotransmitter pathways that play a role in sexual function and dysfunction, providing a theoretical way that THC may alter sexual functioning. These links need to be more clearly studied and elucidated.

ELIGIBILITY:
Inclusion Criteria:

Female ages 18 to 90 years old, agree to fill out questionnaire

Exclusion Criteria:

Male, Female age less than 18 or over 90 years old, decline to fill out questionnaire

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient participants will be asked upon check-in at their ob/gyn office whether they would like to participate in the questionnaire study. Patients will be asked to complete their questionnaire in the exam room of the ob/gyn practice. Patients who choose to voluntarily participate in the study, will be instructed to place their anonymous questionnaire in a provided blank envelope and seal it as to ensure confidentiality, then return their completed questionnaire to the front desk and place the sealed envelope in a lock box themselves.
Sampling Method: Probability Sample
Enrollment: 373 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the relationship between marijuana consumption and sexual function | 1 day
  Study participants will fill out one anonymous questionnaire and deposit the completed questionnaire themselves in a locked box.

CONTACTS AND LOCATIONS:
Overall Officials: Becky Lynn, MD, Principal Investigator — St. Louis University
Locations (1):
- St. Mary's Health Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No